CLINICAL TRIAL: NCT01210352
Title: An Open-Label, Non-randomized, Multicenter, Ascending Dose by Age, Single- and Multiple-Dose Evaluation of the Effectiveness, Safety, and Tolerability of Oral Liquid Oxymorphone HCl Immediate-Release Oral Liquid for Acute Postoperative Pain in Pediatric Subjects
Brief Title: Effectiveness, Safety, and Tolerability Study of Oxymorphone Immediate Release (IR) Oral Liquid in Post Surgical Pediatric Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3319-302
Record Dates: First submitted 2010-09-17; First posted 2010-09-28 (Estimated); Results first posted 2019-05-07 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2019-05

CONDITIONS: Post Operative Pain
Keywords: surgical pain; acute pain; Acute Post Surgical Pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Oxymorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CII Drug (Experimental): Open Label
  Interventions: Drug: oxymorphone HCl

INTERVENTIONS:
Drug: oxymorphone HCl — Comparison of different dosages of drug, 0.05mg/kg, 0.10mg/kg, 0.15mg/kg or 0.20mg/kg oral liquid oxymorphone
  Other Names: Opana

SUMMARY:
The purpose of this study is to evaluate the effectiveness, tolerability, and safety of oxymorphone immediate release (IR) oral liquid as an analgesic for acute postoperative pain in pediatric subjects.

This post marketing study was required by the FDA. Endo Pharmaceuticals Inc. no longer promotes opioids and no longer markets Opana® ER.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 2 to ≤12 years of age. Females of child-bearing potential must be practicing abstinence or using a medically acceptable form of contraception (eg, intrauterine device, hormonal birth control, or double barrier method). For the purpose of this study, all peri- and post-pubertal females will be considered to be of child-bearing potential unless they are biologically sterile or surgically sterile for more than 1 year
2. Subjects must be at least 10 kg and BMI ≤30
3. Scheduled to have a surgery for which oral opioid analgesia will be needed to manage postoperative pain for at least 24 hours (Single-Dose Phase) or 48 hours (Multiple-Dose Phase)following intraoperative and/or postoperative parenteral analgesia
4. Be hospital inpatients, expected to be hospitalized for at least 24 hours (Single-Dose Phase) and 48 hours (Multiple-Dose Phase) following the initial administration of oxymorphone immediate release
5. Available lab results, either intraoperatively (prior to surgical incision) or from within 21 days preoperatively, for clinical chemistry and hematology laboratory analytes (the results must have been reviewed by the Investigator for study eligibility)
6. Able to provide pain assessment evaluations using an age-appropriate instrument provided in the protocol
7. On an intravenous analgesic regimen utilizing a short-acting opioid analgesic following surgery AND anticipated to be switched to an oral opioid as part of the analgesic regimen (according to institution SOC)
8. Demonstrated the ability to tolerate clear fluids following surgery according to the SOC at each institution
9. Informed of the nature of the study and written informed consent has been obtained from the legally responsible parent(s)/legal guardian(s)
10. Provided assent in accordance with IRB requirements
11. Line in place for blood sampling

Exclusion Criteria:

1. Known allergies or sensitivities to oxymorphone or other opioid analgesics
2. Known sensitivity to any component of the study drug
3. Life expectancy <4 weeks
4. Positive pregnancy test at screening (females of reproductive age only)
5. Pregnant and/or lactating
6. Cyanotic heart disease
7. Respiratory, hepatic, renal, neurological, psychological disease, or any other clinically significant condition that would, in the Investigator's opinion, preclude participation in the study
8. Preoperative opioids administered for a period of more than 72 hours in duration
9. Abdominal trauma that would interfere with absorption of study drug
10. Increased intracranial pressure
11. Respiratory condition requiring intubation
12. History of uncontrolled seizures that are not being managed with anticonvulsants
13. Significant prior history of substance abuse or alcohol abuse
14. Received any investigational drug within 30 days prior to the first dose of study drug, or are scheduled to receive an investigational drug other than oxymorphone HCl immediate-release oral liquid during the course of the study
15. Received a monoamine oxidase inhibitor (MAOI) within 14 days prior to the start of study drug
16. Received oxycodone or oxymorphone within 48 hours prior to study start
17. Investigator anticipates that the subject and/or parent(s)/legal guardian(s) would be unable to comply with the protocol
18. Subject (and/or parent[s]/legal guardian[s]) is(are) unable to communicate effectively with study personnel at an age-appropriate level

Ages: 0 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2010-12-13 (Actual); Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saji Vijayan, MD, Study Director — Endo Pharmaceuticals
Locations (8):
- United States (8):
  - Endo Clinical Trial Site #19, Tucson, Arizona
  - Endo Clinical Trial Site #1, Little Rock, Arkansas
  - Endo Clinical Trial Site #3, Aurora, Colorado
  - Endo Clinical Trial Site #6, Indianapolis, Indiana
  - Endo Clinical Trial Site #11, Oklahoma City, Oklahoma
  - Endo Clinical Trial Site #12, Pittsburgh, Pennsylvania
  - Endo Clinical Trial Site #13, Nashville, Tennessee
  - Endo Clinical Trial Site #14, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Dose Phase 6 to ≤12 Years Age Group: 0.05 mg/kg: 6 to ≤12 year age group in the Single Dose Phase given 0.05 mg/kg oxymorphone HCl IR oral liquid
- Single-Dose Phase 6 to ≤12 Years Age Group: 0.10 mg/kg: 6 to ≤12 year age group in the Single Dose Phase given 0.10 mg/kg oxymorphone HCl IR oral liquid
- Single Dose Phase 6 to ≤12 Years Age Group: 0.20 mg/kg: 6 to ≤12 year age group in the Single Dose Phase given 0.20 mg/kg oxymorphone HCl IR oral liquid
- Single Dose Phase 2 to <6 Years Age Group: 0.05 mg/kg: 2 to <6 Years age group in the Single Dose Phase given 0.05 mg/kg oxymorphone HCl IR oral liquid
- Single Dose Phase 2 to <6 Years Age Group: 0.10 mg/kg: 2 to <6 Years age group in the Single Dose Phase given 0.10 mg/kg oxymorphone HCl IR oral liquid
- Single Dose Phase 2 to <6 Years Age Group: 0.20 mg/kg: 2 to <6 Years age group in the Single Dose Phase given 0.20 mg/kg oxymorphone HCl IR oral liquid
- Single Dose Phase 0 to < 2 Years Age Group: 0.05 mg/kg: 0 to < 2 Years age group in the Single Dose Phase given 0.05 mg/kg oxymorphone HCl IR oral liquid
- Multiple Dose Phase 6 to ≤12 Years Age Group: 0.20 mg/kg: 6 to ≤12 year age group in the Multiple Dose Phase given 0.20 mg/kg oxymorphone HCl IR oral liquid
- Multiple Dose Phase 2 to <6 Years Age Group: 0.20 mg/kg: 2 to <6 year age group in the Multiple Dose Phase given 0.20 mg/kg oxymorphone HCl IR oral liquid
Period: Overall Study
Arm/Group | Single Dose Phase 6 to ≤12 Years Age Group: 0.05 mg/kg | Single-Dose Phase 6 to ≤12 Years Age Group: 0.10 mg/kg | Single Dose Phase 6 to ≤12 Years Age Group: 0.20 mg/kg | Single Dose Phase 2 to <6 Years Age Group: 0.05 mg/kg | Single Dose Phase 2 to <6 Years Age Group: 0.10 mg/kg | Single Dose Phase 2 to <6 Years Age Group: 0.20 mg/kg | Single Dose Phase 0 to < 2 Years Age Group: 0.05 mg/kg | Multiple Dose Phase 6 to ≤12 Years Age Group: 0.20 mg/kg | Multiple Dose Phase 2 to <6 Years Age Group: 0.20 mg/kg
Started | 6 | 6 | 7 | 7 | 6 | 6 | 7 | 10 | 6
Completed | 6 | 6 | 5 | 7 | 6 | 6 | 5 | 7 | 2
Not Completed | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Patient Discharged Early | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose Phase 6 to ≤12 Years Age Group: 0.05 mg/kg | Single-Dose Phase 6 to ≤12 Years Age Group: 0.10 mg/kg | Single Dose Phase 6 to ≤12 Years Age Group: 0.20 mg/kg | Single Dose Phase 2 to <6 Years Age Group: 0.05 mg/kg | Single Dose Phase 2 to <6 Years Age Group: 0.10 mg/kg | Single Dose Phase 2 to <6 Years Age Group: 0.20 mg/kg | Single Dose Phase 0 to < 2 Years Age Group: 0.05 mg/kg | Multiple Dose Phase 6 to ≤12 Years Age Group: 0.20 mg/kg | Multiple Dose Phase 2 to <6 Years Age Group: 0.20 mg/kg | Total
Number analyzed (Participants) | 6 | 6 | 7 | 7 | 6 | 6 | 7 | 10 | 6 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.3 (1.75) | 8.7 (1.86) | 9.0 (2.16) | 3.4 (1.27) | 3.5 (1.38) | 3.5 (1.38) | 0.4 (0.53) | 9.6 (1.90) | 3.8 (1.17) | 5.8 (3.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 6 | 2 | 3 | 6 | 1 | 5 | 0 | 26
  Male | 5 | 4 | 1 | 5 | 3 | 0 | 6 | 5 | 6 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 6 | 6 | 6 | 7 | 6 | 4 | 7 | 10 | 6 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 3 | 1 | 0 | 1 | 3 | 1 | 12
  White | 4 | 3 | 6 | 4 | 4 | 6 | 6 | 7 | 5 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 35.25 (11.725) | 30.33 (17.731) | 37.26 (20.613) | 18.76 (4.026) | 15.77 (4.303) | 17.88 (4.869) | 9.10 (3.106) | 41.81 (18.103) | 17.83 (2.701) | 25.84 (16.311)

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Score of Oxymorphone IR Oral Liquid in Pediatric Subjects by Age Group and Time Points in Single Dose Phase
Description: Faces Pain Scale-Revised (FPS-R) was used for the 6 to ≤ 12 years age group, (0 = no pain and 10 = very much pain).
  Face, Legs, Activity, Cry, and Consolability (FLACC) behavior measurement was used for the 2 years to < 6 years and 0 years to < 2 years age groups, (0 = no pain and 10 = very much pain).
Time Frame: Baseline, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post dose; and at the time of rescue
Population: Effectiveness Population. The analyses performed for this study report did not differentiate the pain intensity and pain intensity difference by age/dose combination.
  The analyses were conducted by age group alone and results are presented accordingly.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 6 Years to ≤ 12 Years Age Group in Single Dose Phase: Faces Pain Scale-Revised (FPS-R) was used for the 6 to ≤ 12 years age group
- 2 Years to < 6 Years Age Group in Single Dose Phase: Face, Legs, Activity, Cry, and Consolability (FLACC) behavior measurement was used for the 2 years to < 6 year age group
- 0 Years to < 2 Years Age Group in Single Dose Phase: Face, Legs, Activity, Cry, and Consolability (FLACC) behavior measurement was used for the 0 years to < 2 years age group
Arm/Group | 6 Years to ≤ 12 Years Age Group in Single Dose Phase | 2 Years to < 6 Years Age Group in Single Dose Phase | 0 Years to < 2 Years Age Group in Single Dose Phase
Number analyzed (Participants) | 19 | 19 | 7
score on a scale
  Baseline (Prior to Treatment) | 4.5 (3.12) | 3.4 (3.55) | 2.4 (1.90)
  15 Minutes Post Dose: number analyzed (Participants) | 19 | 18 | 7
  15 Minutes Post Dose | 3.5 (3.64) | 1.2 (2.50) | 1.3 (2.63)
  30 Minutes Post Dose: number analyzed (Participants) | 18 | 18 | 7
  30 Minutes Post Dose | 2.7 (3.29) | 1.2 (2.28) | 0.4 (0.79)
  1 Hour Post Dose: number analyzed (Participants) | 18 | 17 | 7
  1 Hour Post Dose | 1.8 (1.93) | 0.2 (0.56) | 0.1 (0.38)
  1.5 Hours Post Dose: number analyzed (Participants) | 12 | 11 | 0
  1.5 Hours Post Dose | 2.0 (2.56) | 0.2 (0.60) |
  2 Hours Post Dose: number analyzed (Participants) | 15 | 16 | 7
  2 Hours Post Dose | 3.1 (3.37) | 0.4 (0.81) | 0.4 (0.79)
  3 Hours Post Dose: number analyzed (Participants) | 4 | 3 | 7
  3 Hours Post Dose | 0.0 (0.00) | 2.0 (2.65) | 0.4 (1.13)
  4 Hours Post Dose: number analyzed (Participants) | 12 | 11 | 6
  4 Hours Post Dose | 1.8 (2.17) | 1.5 (2.34) | 1.3 (1.51)
  6 Hours Post Dose: number analyzed (Participants) | 7 | 9 | 4
  6 Hours Post Dose | 2.3 (1.80) | 0.7 (1.41) | 0.8 (1.50)
  8 Hours Post Dose: number analyzed (Participants) | 3 | 8 | 3
  8 Hours Post Dose | 3.3 (5.77) | 0.8 (1.39) | 0.0 (0.00)
  12 Hours Post Dose: number analyzed (Participants) | 3 | 6 | 3
  12 Hours Post Dose | 1.3 (2.31) | 0.0 (0.00) | 0.0 (0.00)
  24 Hours Post Dose: number analyzed (Participants) | 0 | 4 | 2
  24 Hours Post Dose |  | 0.0 (0.00) | 0.0 (0.00)

2. Primary Outcome: Descriptive Statistics of the Pain Intensity Difference (PID) by Age Group and Time Points in Single-Dose Phase
Description: Faces Pain Scale-Revised (FPS-R) was used for the 6 to ≤ 12 years age group, (0 = no pain and 10 = very much pain).
  Face, Legs, Activity, Cry, and Consolability (FLACC) behavior measurement was used for the 2 years to < 6 years and 0 years to < 2 years age groups, (0 = no pain and 10 = very much pain).
  PID was calculated as the pain intensity score at baseline minus the current pain intensity score at each corresponding time point.
Time Frame: Baseline (prior to dose); 15, 30 minutes, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours post-dose; and at the time of rescue
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 0 Years to < 2 Years Age Group in Single Dose Phase: Face, Legs, Activity, Cry, and Consolability (FLACC) behavior measurement was used for the 0 years to < 2 year age group
Arm/Group | 6 Years to ≤ 12 Years Age Group in Single Dose Phase | 2 Years to < 6 Years Age Group in Single Dose Phase | 0 Years to < 2 Years Age Group in Single Dose Phase
Number analyzed (Participants) | 19 | 19 | 7
score on a scale
  15 Minutes Post-Dose: number analyzed (Participants) | 19 | 18 | 7
  15 Minutes Post-Dose | 1.1 (4.24) | 2.1 (2.56) | 1.1 (4.06)
  30 Minutes Post-Dose: number analyzed (Participants) | 18 | 18 | 7
  30 Minutes Post-Dose | 1.6 (3.33) | 2.1 (2.49) | 2.0 (2.45)
  1 Hour Post-Dose: number analyzed (Participants) | 18 | 17 | 7
  1 Hour Post-Dose | 2.4 (3.67) | 2.6 (3.10) | 2.3 (1.98)
  1.5 Hours Post-Dose: number analyzed (Participants) | 12 | 11 | 0
  1.5 Hours Post-Dose | 3.0 (3.86) | 3.8 (3.84) |
  2 Hours Post-Dose: number analyzed (Participants) | 15 | 16 | 7
  2 Hours Post-Dose | 1.5 (4.03) | 2.6 (3.40) | 2.0 (2.45)
  3 Hours Post-Dose: number analyzed (Participants) | 4 | 3 | 7
  3 Hours Post-Dose | 3.0 (2.00) | -1.0 (2.00) | 2.0 (2.31)
  4 Hours Post-Dose: number analyzed (Participants) | 12 | 11 | 6
  4 Hours Post-Dose | 2.7 (4.21) | 2.5 (3.24) | 1.0 (2.83)
  6 Hours Post-Dose: number analyzed (Participants) | 7 | 9 | 4
  6 Hours Post-Dose | 3.1 (4.14) | 3.0 (2.40) | 1.0 (2.71)
  8 Hours Post-Dose: number analyzed (Participants) | 3 | 8 | 3
  8 Hours Post-Dose | 1.3 (2.31) | 2.4 (2.92) | 1.7 (2.89)
  12 Hours Post-Dose: number analyzed (Participants) | 3 | 6 | 3
  12 Hours Post-Dose | 3.3 (5.77) | 3.2 (2.32) | 1.7 (2.89)
  24 Hours Post-Dose: number analyzed (Participants) | 0 | 4 | 2
  24 Hours Post-Dose |  | 3.0 (2.16) | 0.0 (0.00)

3. Primary Outcome: Pain Intensity Score of Oxymorphone IR Oral Liquid in Pediatric Subjects by Age Group and Time Points in Multiple Dose Phase
Description: as for outcome 1
Time Frame: Baseline, 0.5, 1, 1.5, 2, hours post dose, and immediately prior to all remaining doses administered through 48 hours after administration of the initial dose; and at time of rescue
Population: Effectiveness Population. Based on the recommendation of the Independent Data Monitoring Committee (IDMC), there was only 1 dose group of 0.2 mg/kg administered during the Multiple-dose Phase. Thus, this outcome measure was only assessed in this dose group.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 6 Years to ≤ 12 Years Age Group in Multiple Dose Phase: Faces Pain Scale-Revised (FPS-R) was used for the 6 to ≤ 12 years age group
- 2 Years to < 6 Years Age Group in Multiple Dose Phase: Face, Legs, Activity, Cry, and Consolability (FLACC) behavior measurement was used for the 2 years to < 6 year age group
Arm/Group | 6 Years to ≤ 12 Years Age Group in Multiple Dose Phase | 2 Years to < 6 Years Age Group in Multiple Dose Phase
Number analyzed (Participants) | 10 | 6
score on a scale
  Dose 1, Baseline (Prior to Treatment): number analyzed (Participants) | 9 | 6
  Dose 1, Baseline (Prior to Treatment) | 3.1 (2.67) | 3.5 (3.27)
  Dose 1, 30 Minutes Post Dose: number analyzed (Participants) | 9 | 6
  Dose 1, 30 Minutes Post Dose | 2.7 (1.73) | 1.3 (1.97)
  Dose 1, 1 Hour Post Dose: number analyzed (Participants) | 10 | 5
  Dose 1, 1 Hour Post Dose | 2.0 (2.83) | 1.8 (2.05)
  Dose 1, 1.5 Hours Post Dose: number analyzed (Participants) | 8 | 4
  Dose 1, 1.5 Hours Post Dose | 2.3 (1.67) | 0.0 (0.00)
  Dose 1, 2 Hours Post Dose: number analyzed (Participants) | 8 | 4
  Dose 1, 2 Hours Post Dose | 2.8 (2.38) | 0.0 (0.00)
  Dose 2, 0 Hour: number analyzed (Participants) | 7 | 3
  Dose 2, 0 Hour | 4.0 (3.27) | 5.0 (2.65)
  Dose 3, 0 Hour: number analyzed (Participants) | 5 | 3
  Dose 3, 0 Hour | 5.6 (2.61) | 3.7 (3.21)
  Dose 4, 0 Hour: number analyzed (Participants) | 6 | 2
  Dose 4, 0 Hour | 4.0 (3.58) | 4.5 (0.71)
  Dose 5, 0 Hour: number analyzed (Participants) | 4 | 2
  Dose 5, 0 Hour | 2.5 (1.00) | 5.0 (0.00)
  Dose 6, 0 Hour: number analyzed (Participants) | 4 | 1
  Dose 6, 0 Hour | 2.5 (1.00) | 6.0 (NA) — SD cannot be derived based on one subject data point
  Dose 7, 0 Hour: number analyzed (Participants) | 4 | 0
  Dose 7, 0 Hour | 3.0 (2.00) |
  Dose 8, 0 Hour: number analyzed (Participants) | 3 | 0
  Dose 8, 0 Hour | 4.7 (2.31) |
  Dose 9, 0 Hour: number analyzed (Participants) | 3 | 0
  Dose 9, 0 Hour | 1.3 (1.15) |
  Dose 10, 0 Hour: number analyzed (Participants) | 3 | 0
  Dose 10, 0 Hour | 2.0 (0.00) |
  Dose 11, 0 Hour: number analyzed (Participants) | 2 | 0
  Dose 11, 0 Hour | 2.0 (0.00) |
  Dose 12, 0 Hour: number analyzed (Participants) | 2 | 0
  Dose 12, 0 Hour | 5.0 (4.24) |
  End of Study/Early Termination: number analyzed (Participants) | 4 | 4
  End of Study/Early Termination | 4.0 (1.63) | 1.3 (2.50)

4. Primary Outcome: Descriptive Statistics of Pain Intensity Difference (PID) by Age Group and Time Points in Multiple-Dose Phase
Description: Faces Pain Scale-Revised (FPS-R) was used for the 6 to ≤ 12 years age group, (0 = no pain and 10 = very much pain).
  Face, Legs, Activity, Cry, and Consolability (FLACC) behavior measurement was used for the 2 years to < 6 years and 0 years to < 2 years age groups, (0 = no pain and 10 = very much pain).
  PID is calculated as the pain intensity score at baseline minus the current pain intensity score at each corresponding time point.
Time Frame: 0.5, 1, 1.5, 2, hours post dose 1 through to Dose 12, 0 Hour; End of Study/Early Termination
Population: Effectiveness Population.IDMC recommended dose: 0.20 mg/kg oxymorphone HCl oral solution for the Multiple-dose Phase. Therefore, the analyses were conducted in a total of 16 subjects ranging from 2 to ≤12 years who received the dose of 0.20 mg/kg oxymorphone HCl oral solution as shown in the table of baseline characteristic in the participant flow.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- 6 to ≤12 Years Age Group: 0.20 mg/kg: Faces Pain Scale-Revised (FPS-R) was used for the 6 to ≤ 12 years age group
- 2 to <6 Years Age Group: 0.20 mg/kg: Face, Legs, Activity, Cry, and Consolability (FLACC) behavior measurement was used for the 2 years to < 6 year age group
Arm/Group | 6 to ≤12 Years Age Group: 0.20 mg/kg | 2 to <6 Years Age Group: 0.20 mg/kg
Number analyzed (Participants) | 10 | 6
score on a scale
  Dose 1, 30 Minutes Post-Dose: number analyzed (Participants) | 9 | 6
  Dose 1, 30 Minutes Post-Dose | 0.4 (2.19) | 2.2 (2.79)
  Dose 1, 1 Hour Post-Dose: number analyzed (Participants) | 9 | 5
  Dose 1, 1 Hour Post-Dose | 0.9 (2.67) | 2.0 (3.46)
  Dose 1, 1.5 Hours Post-Dose: number analyzed (Participants) | 7 | 4
  Dose 1, 1.5 Hours Post-Dose | 1.1 (3.02) | 4.8 (3.30)
  Dose 1, 2 Hours Post-Dose: number analyzed (Participants) | 8 | 4
  Dose 1, 2 Hours Post-Dose | 0.0 (1.85) | 4.8 (3.30)
  Dose 2, 0 Hour: number analyzed (Participants) | 6 | 3
  Dose 2, 0 Hour | -2.3 (3.88) | 0.3 (1.53)
  Dose 3, 0 Hour: number analyzed (Participants) | 4 | 3
  Dose 3, 0 Hour | -3.5 (4.43) | 1.7 (0.58)
  Dose 4, 0 Hour: number analyzed (Participants) | 5 | 2
  Dose 4, 0 Hour | -0.8 (3.03) | 3.0 (1.41)
  Dose 5, 0 Hour: number analyzed (Participants) | 4 | 2
  Dose 5, 0 Hour | 1.0 (1.15) | 2.5 (0.71)
  Dose 6, 0 Hour: number analyzed (Participants) | 4 | 1
  Dose 6, 0 Hour | 1.0 (2.58) | 2.0 (NA) — Not determined, or not reported due to insufficient data for reliable estimate
  Dose 7, 0 Hour: number analyzed (Participants) | 4 | 0
  Dose 7, 0 Hour | 0.5 (2.52) |
  Dose 8, 0 Hour: number analyzed (Participants) | 3 | 0
  Dose 8, 0 Hour | -2.0 (2.00) |
  Dose 9, 0 Hour: number analyzed (Participants) | 3 | 0
  Dose 9, 0 Hour | 2.7 (1.15) |
  Dose 10, 0 Hour: number analyzed (Participants) | 3 | 0
  Dose 10, 0 Hour | 2.0 (2.00) |
  Dose 11, 0 Hour: number analyzed (Participants) | 2 | 0
  Dose 11, 0 Hour | 3.0 (1.41) |
  Dose 12, 0 Hour: number analyzed (Participants) | 2 | 0
  Dose 12, 0 Hour | 0.0 (5.66) |
  End of Study/Early Termination: number analyzed (Participants) | 4 | 4
  End of Study/Early Termination | -0.5 (1.91) | 3.5 (3.11)

5. Primary Outcome: Number (%) of Subjects With Rescue Medication Use by Age and Dose Group in Multiple-Dose Phase
Description: Rescue Medication Use in Multiple Dose Phase
Time Frame: Rescue Medication Use
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Groups:
- 6 to ≤12 Years Age Group: 0.20 mg/kg; 2 to <6 Years Age Group: 0.20 mg/kg: Percentages are based on the number of subjects ('N') in effectiveness population in each dose group in each age group in Multiple-Dose Phase
Arm/Group | 6 to ≤12 Years Age Group: 0.20 mg/kg | 2 to <6 Years Age Group: 0.20 mg/kg
Number analyzed (Participants) | 10 | 6
Participants
  Rescue Medication Used | 5 | 2
  No Rescue Medication needed | 5 | 4

6. Secondary Outcome: Oxymorphone Cmax Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: Cmax: Maximum plasma concentration; the highest concentration observed during a dosage interval
Time Frame: Serial blood samples were collected at time 0 (Baseline), at 15 and 30 minutes, and at 1, 1.5, 2, 4, 6, 8, 12, and 24 hours post-dose
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose: Cmax: Maximum plasma concentration; the highest concentration observed during a dosage interval
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 7 | 6
ng/mL | 0.415 (0.211) | 0.33 (0.217) | 1.14 (0.847) | 1.76 (1.62) | 1.33 (0.772) | 3.16 (1.65)

7. Secondary Outcome: Oxymorphone Tmax Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: Tmax: The time at which Cmax was observed
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h
Groups:
- 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose: Tmax: The time at which Cmax was observed
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 7 | 6
h | 2.7 (1.66) | 2.64 (1.03) | 1.38 (1.3) | 1.45 (1.39) | 2.49 (3.17) | 1.59 (1.38)

8. Secondary Outcome: Oxymorphone Clast Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: Clast: Minimum plasma concentration; the last concentration observed during a dosage interval
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose: Clast: Minimum plasma concentration; the last concentration observed during a dosage interval
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 7 | 6
ng/mL | 0.0759 (0.072) | 0.0618 (0.0389) | 0.11 (0.0847) | 0.0671 (0.0376) | 0.269 (0.182) | 0.645 (1.3)

9. Secondary Outcome: Oxymorphone Tlast Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: Tlast: The time at which Clast was observed
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h
Groups:
- 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose: Tlast: The time at which Clast was observed
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 7 | 6
h | 15.4 (7.01) | 13.2 (5.06) | 18 (6.55) | 16 (8.04) | 12.6 (9.85) | 18.4 (8.97)

10. Secondary Outcome: Oxymorphone AUC0-t Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: AUC0-t: Area under the concentration versus time curve from time 0 to the last measured concentration (Clast) calculated by linear trapezoidal rule
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose: AUC0-t: Area under the concentration versus time curve from time 0 to the last measured concentration (Clast) calculated by linear trapezoidal rule
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 7 | 6
h*ng/mL | 2.56 (2) | 1.69 (0.943) | 3.01 (0.766) | 3.99 (2.09) | 5.32 (4.53) | 9.37 (5.81)

11. Secondary Outcome: Oxymorphone AUC0-inf Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: AUC0-inf: Area under the concentration versus time curve from time 0 to infinity, calculated as AUC0-t + Clast/λn
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose: AUC0-inf: Area under the concentration versus time curve from time 0 to infinity, calculated as AUC0-t + Clast/λn
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 3 | 2
h*ng/mL | NA (0.0516) — Not determined, or not reported due to insufficient data for reliable estimate | 3.22 (1.56) | 3.01 (0.946) | 3.69 (3.12) | 6.92 (4.02) | 14.3 (5.01)

12. Secondary Outcome: Oxymorphone AUC0-24 Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: AUC0-24: Area under the concentration versus time curve from time 0 to 24 hours calculated by linear trapezoidal rule
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose: AUC0-24: Area under the concentration versus time curve from time 0 to 24 hours calculated by linear trapezoidal rule
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 3 | 3 | 4 | 4 | 4 | 2
h*ng/mL | 3.75 (2.32) | 2.65 (1.4) | 3.01 (0.905) | 3.69 (2.44) | 6.11 (2.83) | 14 (4.72)

13. Secondary Outcome: Oxymorphone t1/2 Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: t1/2: Terminal half-life, calculated as λn/(ln 2)
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h
Groups:
- 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose; 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose: t1/2: Terminal half-life, calculated as λn/(ln 2)
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 2 | 2 | 2 | 3 | 3 | 2
h | NA (0.232) — Not determined, or not reported due to insufficient data for reliable estimate | 5.01 (1.4) | 7.5 (7.33) | 4.38 (2.9) | 5.13 (3.16) | 4.39 (1.16)

14. Secondary Outcome: Dose-Normalized Oxymorphone CL/F Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: CL/F: Apparent oral clearance, calculated as Dose/AUC0-inf
Time Frame: as for outcome 6
Population: PK Population (subjects with sufficient plasma concentration data to calculate PK parameter values). Since the overall exposure (AUC 0 to t) increased in near dose proportional manner, PK parameter values were dose normalized across all dose levels for each age group to determine the CL/F.
Measure: Mean (Standard Deviation); unit: L/h/kg
Groups:
- Combined 0.05, 0.1, and 0.2 mg/kg - Aged 6 Years to ≤ 12 Years; Combined 0.05, 0.1, and 0.2 mg/kg - Aged 2 Years to <6 Years: CL/F: Apparent oral clearance, calculated as Dose/AUC0-inf
Arm/Group | Combined 0.05, 0.1, and 0.2 mg/kg - Aged 6 Years to ≤ 12 Years | Combined 0.05, 0.1, and 0.2 mg/kg - Aged 2 Years to <6 Years
Number analyzed (Participants) | 7 | 7
L/h/kg | 31.2 (13.6) | 26.4 (18.8)

15. Secondary Outcome: Dose-Normalized Oxymorphone V/F Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: V/F: Apparent volume of distribution, calculated as Dose/(AUC0-inf * λn)
Time Frame: as for outcome 6
Population: PK Population (subjects with sufficient plasma concentration data to calculate PK parameter values). Since the overall exposure (AUC 0 to t) increased in near dose proportional manner, PK parameter values were dose normalized across all dose levels for each age group to determine the V/F.
Measure: Mean (Standard Deviation); unit: L/kg
Groups:
- Combined 0.05, 0.1, and 0.2 mg/kg - Aged 6 Years to ≤ 12 Years; Combined 0.05, 0.1, and 0.2 mg/kg - Aged 2 Years to <6 Years: V/F: Apparent volume of distribution, calculated as Dose/(AUC0-inf * λn)
Arm/Group | Combined 0.05, 0.1, and 0.2 mg/kg - Aged 6 Years to ≤ 12 Years | Combined 0.05, 0.1, and 0.2 mg/kg - Aged 2 Years to <6 Years
Number analyzed (Participants) | 7 | 7
L/kg | 205 (145) | 154 (121)

16. Secondary Outcome: Oxymorphone Cmax Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: Cmax: Maximum plasma concentration; the highest concentration observed during a dosage interval
Time Frame: Serial blood samples were collected at: time 0 (Baseline), at 0.5, 1, 1.5, and 2 hours post-Dose 1, immediately prior to Doses 2, 3, 4, 5, 6, 7, and at 0.5, 1, 1.5, and 2 hours post-Dose 7
Population: Analysis was conducted in the PK Population with sufficient concentration data at required time points. During the Multiple-dose Phase, all subjects received 0.2 mg/kg oxymorphone HCl IR solution. Analysis of Cmax was conducted in the subjects remaining in the study, with sufficient concentration data at the required time points, as shown.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7: Cmax: Maximum plasma concentration; the highest concentration observed during a dosage interval
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 10 | 5 | 3 | 0
ng/mL | 1.46 (1.16) | 2.58 (1.24) | 2.66 (0.805) |

17. Secondary Outcome: Oxymorphone Tmax Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: Tmax: The time at which Cmax was observed
Time Frame: as for outcome 16
Population: Analysis was conducted in the PK Population with sufficient concentration data at required time points. During the Multiple-dose Phase, all subjects received 0.2 mg/kg oxymorphone HCl IR solution. Analysis of Tmax was conducted in the subjects remaining in the study, with sufficient concentration data at the required time points, as shown.
Measure: Mean (Standard Deviation); unit: h
Groups:
- 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7: Tmax: The time at which Cmax was observed
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 10 | 5 | 3 | 0
h | 1.37 (0.599) | 0.967 (0.622) | 1.21 (1.1) |

18. Secondary Outcome: Oxymorphone Clast Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: Clast: Minimum plasma concentration; the last concentration observed during a dosage interval
Time Frame: as for outcome 16
Population: Analysis was conducted in the PK Population with sufficient concentration data at required time points. During the Multiple-dose Phase, all subjects received 0.2 mg/kg oxymorphone HCl IR solution. Analysis of Clast was conducted in the subjects remaining in the study, with sufficient concentration data at the required time points, as shown.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7: Clast: Minimum plasma concentration; the last concentration observed during a dosage interval
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 10 | 5 | 3 | 0
ng/mL | 0.452 (0.286) | 0.508 (0.32) | 2.3 (0.745) |

19. Secondary Outcome: Oxymorphone Tlast Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: Tlast: The time at which Clast was observed
Time Frame: as for outcome 16
Population: Analysis was conducted in the PK Population with sufficient concentration data at required time points. During the Multiple-dose Phase, all subjects received 0.2 mg/kg oxymorphone HCl IR solution. Analysis of Tlast was conducted in the subjects remaining in the study, with sufficient concentration data at the required time points, as shown.
Measure: Mean (Standard Deviation); unit: h
Groups:
- 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7: Tlast: The time at which Clast was observed
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 10 | 5 | 3 | 0
h | 4 (0.971) | 4.47 (1.68) | 2.09 (0.077) |

20. Secondary Outcome: Oxymorphone AUC0-t Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: as for outcome 10
Time Frame: as for outcome 16
Population: Analysis was conducted in the PK Population with sufficient concentration data at required time points. During the Multiple-dose Phase, all subjects received 0.2 mg/kg oxymorphone HCl IR solution. Analysis of AUC0-t was conducted in the subjects remaining in the study, with sufficient concentration data at the required time points, as shown.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7: AUC0-t: Area under the concentration versus time curve from time 0 to the last measured concentration (Clast) calculated by linear trapezoidal rule
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 10 | 5 | 3 | 0
h*ng/mL | 3.49 (3.22) | 3.88 (1.45) | 4.24 (0.9) |

21. Secondary Outcome: Oxymorphone AUC0-inf Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: AUC0-inf: Area under the concentration versus time curve from time 0 to infinity, calculated as AUC0-t + Clast/λn
Time Frame: as for outcome 16
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7: AUC0-inf: Area under the concentration versus time curve from time 0 to infinity, calculated as AUC0-t + Clast/λn
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 3 | 3 | 0 | 0
h*ng/mL | 4.01 (1.43) | 4.53 (2.21) |  |

22. Secondary Outcome: Oxymorphone AUC0-24 Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: AUC0-24: Area under the concentration versus time curve from time 0 to 24 hours calculated by linear trapezoidal rule
Time Frame: as for outcome 16
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7: AUC0-24: Area under the concentration versus time curve from time 0 to 24 hours calculated by linear trapezoidal rule
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 3 | 3 | 0 | 0
h*ng/mL | 4.01 (1.42) | 4.53 (2.21) |  |

23. Secondary Outcome: Oxymorphone t1/2 Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: t1/2: Terminal half-life, calculated as λn/(ln 2)
Time Frame: as for outcome 16
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h
Groups:
- 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1; 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7; 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7: t1/2: Terminal half-life, calculated as λn/(ln 2)
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 3 | 3 | 0 | 0
h | 2.18 (0.459) | 1.17 (0.632) |  |

24. Secondary Outcome: 6 Beta-Hydroxyoxymorphone Cmax Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: Cmax: Maximum plasma concentration; the highest concentration observed during a dosage interval
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 7 | 6
ng/mL | 0.104 (0.0555) | 0.1 (0.073) | 0.384 (0.177) | 0.437 (0.419) | 0.603 (0.513) | 0.587 (0.182)

25. Secondary Outcome: 6 Beta-Hydroxyoxymorphone Tmax Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: Tmax: The time at which Cmax was observed
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 7 | 6
h | 2.86 (1.17) | 2.91 (1.11) | 1.38 (1.3) | 1.86 (1.69) | 3.08 (3.42) | 1.93 (1.71)

26. Secondary Outcome: 6 Beta-Hydroxyoxymorphone Clast Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: Clast: Minimum plasma concentration; the last concentration observed during a dosage interval
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 7 | 6
ng/mL | 0.0453 (0.0272) | 0.0418 (0.0152) | 0.0568 (0.0292) | 0.0332 (0.0183) | 0.204 (0.188) | 0.0994 (0.144)

27. Secondary Outcome: 6 Beta-Hydroxyoxymorphone Tlast Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: Tlast: The time at which Clast was observed
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 5 | 7 | 6 | 6 | 7 | 6
h | 9.66 (8.25) | 8.86 (7.82) | 14.4 (7.86) | 16.1 (9.05) | 12.6 (9.85) | 18.4 (8.97)

28. Secondary Outcome: 6 Beta-Hydroxyoxymorphone AUC0-t Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: as for outcome 10
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 6 | 7 | 6 | 6 | 7 | 6
h*ng/mL | 0.459 (0.396) | 0.467 (0.473) | 1.22 (0.761) | 1.27 (0.637) | 2.64 (2.52) | 2.26 (1.07)

29. Secondary Outcome: 6 Beta-Hydroxyoxymorphone AUC0-inf Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: AUC0-inf: Area under the concentration versus time curve from time 0 to infinity, calculated as AUC0-t + Clast/λn
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 2 | 2
h*ng/mL | 1.83 (NA) — Not determined, or not reported due to insufficient data for reliable estimate | 1.11 (NA) — Not determined, or not reported due to insufficient data for reliable estimate | 0.535 (NA) — Not determined, or not reported due to insufficient data for reliable estimate | 1.76 (0.762) | 7.58 (5.12) | 2.76 (0.399)

30. Secondary Outcome: 6 Beta-Hydroxyoxymorphone AUC0-24 Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: AUC0-24: Area under the concentration versus time curve from time 0 to 24 hours calculated by linear trapezoidal rule
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 1 | 1 | 3 | 5 | 4 | 2
h*ng/mL | 1.09 (NA) — Not determined, or not reported due to insufficient data for reliable estimate | 1.09 (NA) — Not determined, or not reported due to insufficient data for reliable estimate | 1.08 (0.484) | 1.45 (0.588) | 3.08 (1.32) | 2.61 (0.226)

31. Secondary Outcome: 6 Beta-Hydroxyoxymorphone t1/2 Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: t1/2: Terminal half-life, calculated as λn/(ln 2)
Time Frame: as for outcome 6
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 0.05 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.05 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.1 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.1 mg/kg - Children Aged 2 Years to <6 Years in Single Dose | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years in Single Dose | 0.2 mg/kg - Children Aged 2 Years to <6 Years in Single Dose
Number analyzed (Participants) | 1 | 1 | 1 | 4 | 2 | 2
h | 20.5 (NA) — Not determined, or not reported due to insufficient data for reliable estimate | 4.48 (NA) — Not determined, or not reported due to insufficient data for reliable estimate | 2.31 (NA) — Not determined, or not reported due to insufficient data for reliable estimate | 8.67 (8.06) | 18.7 (22.5) | 5.18 (2.55)

32. Secondary Outcome: Dose-Normalized 6 Beta-Hydroxyoxymorphone CL/F Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: CL/F: Apparent oral clearance, calculated as Dose/AUC0-inf
Time Frame: as for outcome 6
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | Combined 0.05, 0.1, and 0.2 mg/kg - Aged 6 Years to ≤ 12 Years | Combined 0.05, 0.1, and 0.2 mg/kg - Aged 2 Years to <6 Years
Number analyzed (Participants) | 4 | 7
L/h/kg | 70.7 (78.8) | 65 (23.2)

33. Secondary Outcome: Dose-Normalized 6 Beta-Hydroxyoxymorphone V/F Following Single-Dose Administration of 0.05, 0.1, and 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Single-Dose Phase
Description: V/F: Apparent volume of distribution, calculated as Dose/(AUC0-inf * λn)
Time Frame: as for outcome 6
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Combined 0.05, 0.1, and 0.2 mg/kg - Aged 6 Years to ≤ 12 Years | Combined 0.05, 0.1, and 0.2 mg/kg - Aged 2 Years to <6 Years
Number analyzed (Participants) | 4 | 7
L/kg | 631 (308) | 575 (487)

34. Secondary Outcome: 6 Beta-Hydroxyoxymorphone Cmax Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: Cmax: Maximum plasma concentration; the highest concentration observed during a dosage interval
Time Frame: as for outcome 16
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 10 | 5 | 3 | 0
ng/mL | 0.547 (0.472) | 0.829 (0.541) | 1.41 (0.473) |

35. Secondary Outcome: 6 Beta-Hydroxyoxymorphone Tmax Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: Tmax: The time at which Cmax was observed
Time Frame: as for outcome 16
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 10 | 5 | 3 | 0
h | 1.67 (1.01) | 1.37 (1.5) | 1.36 (0.85) |

36. Secondary Outcome: 6 Beta-Hydroxyoxymorphone Clast Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: Clast: Minimum plasma concentration; the last concentration observed during a dosage interval
Time Frame: as for outcome 16
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 10 | 5 | 3 | 0
ng/mL | 0.201 (0.118) | 0.225 (0.139) | 1.25 (0.585) |

37. Secondary Outcome: 6 Beta-Hydroxyoxymorphone Tlast Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: Tlast: The time at which Clast was observed
Time Frame: as for outcome 16
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 10 | 5 | 3 | 0
h | 3.97 (1.05) | 4.47 (1.68) | 2.09 (0.077) |

38. Secondary Outcome: 6 Beta-Hydroxyoxymorphone AUC0-t Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: as for outcome 10
Time Frame: as for outcome 16
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 10 | 5 | 3 | 0
h*ng/mL | 1.35 (1.27) | 1.61 (1.19) | 2.25 (0.547) |

39. Secondary Outcome: 6 Beta-Hydroxyoxymorphone AUC0-inf Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: AUC0-inf: Area under the concentration versus time curve from time 0 to infinity, calculated as AUC0-t + Clast/λn
Time Frame: as for outcome 16
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 3 | 3 | 1 | 0
h*ng/mL | 2.15 (0.769) | 1.79 (1.73) | 7.66 (NA) — Not determined, or not reported due to insufficient data for reliable estimate |

40. Secondary Outcome: 6 Beta-Hydroxyoxymorphone AUC0-24 Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: AUC0-24: Area under the concentration versus time curve from time 0 to 24 hours calculated by linear trapezoidal rule
Time Frame: as for outcome 16
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 3 | 3 | 1 | 0
h*ng/mL | 2.11 (0.748) | 1.78 (1.72) | 7.38 (NA) — Not determined, or not reported due to insufficient data for reliable estimate |

41. Secondary Outcome: 6 Beta-Hydroxyoxymorphone t1/2 Following Multiple-Dose Administration of 0.2 mg/kg Oxymorphone HCl Immediate-Release Oral Liquid in Children Aged 2 Years to ≤12 Years in the Multiple-Dose Phase From Dose 1 and Dose 7
Description: t1/2: Terminal half-life, calculated as λn/(ln 2)
Time Frame: as for outcome 16
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: h
Arm/Group | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 1 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 1 | 0.2 mg/kg - Children Aged 6 Years to ≤12 Years - Dose 7 | 0.2 mg/kg - Children Aged 2 Years to <6 Years - Dose 7
Number analyzed (Participants) | 3 | 3 | 1 | 0
h | 3.61 (1.67) | 1.42 (0.73) | 4.9 (NA) — Not determined, or not reported due to insufficient data for reliable estimate |

ADVERSE EVENTS:
Time Frame: All Single and Multiple Dose Phase (serious and nonserious) AEs, whether elicited during study visits or spontaneously reported by the subject, included events that occurred from the time the subject signed the study-specific ICF until completion of, or discharge from the study.
Description: AEs were recorded from screening visit, throughout the study, until follow-up visit. All AE's were followed until resolved, or for 30 days after the last dose of study medication if the AE remained unresolved or premature discontinuation from the study whether or not related to the investigational product.
Groups:
- 6 Years to ≤ 12 Years Age Group: Single Dose 0.05 mg/kg: All (serious and nonserious) AEs for the 6 years to ≤ 12 years Age Group - Single Dose 0.05 mg/kg
- 6 Years to ≤ 12 Years Age Group: Single Dose 0.10 mg/kg: All (serious and nonserious) AEs for the 6 years to ≤ 12 years Age Group - Single Dose 0.10 mg/kg
- 6 Years to ≤ 12 Years Age Group: Single Dose 0.20 mg/kg: All (serious and nonserious) AEs for the 6 years to ≤ 12 years Age Group - Single Dose 0.20 mg/kg
- 2 Years to < 6 Years Age Group: Single Dose 0.05 mg/kg: All (serious and nonserious) AEs for the 2 years to < 6 years Age Group - Single Dose 0.05 mg/kg
- 2 Years to < 6 Years Age Group: Single Dose 0.10 mg/kg: All (serious and nonserious) AEs for the 2 years to < 6 years Age Group - Single Dose 0.10 mg/kg
- 2 Years to < 6 Years Age Group: Single Dose 0.20 mg/kg: All (serious and nonserious) AEs for the 2 years to < 6 years Age Group - Single Dose 0.20 mg/kg
- 0 to < 2 Years Age Group: Single Dose 0.05 mg/kg: All (serious and nonserious) AEs for the 0 to < 2 years Age Group - Single Dose 0.05 mg/kg
- 6 Years to ≤ 12 Years Age Group: Multiple Dose 0.20 mg/kg: All (serious and nonserious) AEs for the 0 to < 2 years Age Group - Multiple Dose 0.20 mg/kg
- 2 Years to < 6 Years Age Group: Multiple Dose 0.20 mg/kg: All (serious and nonserious) AEs for the 2 to < 6 years Age Group - Multiple Dose 0.20 mg/kg
Arm/Group | 6 Years to ≤ 12 Years Age Group: Single Dose 0.05 mg/kg | 6 Years to ≤ 12 Years Age Group: Single Dose 0.10 mg/kg | 6 Years to ≤ 12 Years Age Group: Single Dose 0.20 mg/kg | 2 Years to < 6 Years Age Group: Single Dose 0.05 mg/kg | 2 Years to < 6 Years Age Group: Single Dose 0.10 mg/kg | 2 Years to < 6 Years Age Group: Single Dose 0.20 mg/kg | 0 to < 2 Years Age Group: Single Dose 0.05 mg/kg | 6 Years to ≤ 12 Years Age Group: Multiple Dose 0.20 mg/kg | 2 Years to < 6 Years Age Group: Multiple Dose 0.20 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/7 | 0/6 | 0/6 | 0/7 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/6 | 0/7 | 1/7 | 0/6 | 0/6 | 0/7 | 2/10 | 0/6
Other Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 4/7 | 7/7 | 5/6 | 3/6 | 4/7 | 10/10 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 6 Years to ≤ 12 Years Age Group: Single Dose 0.05 mg/kg (N=6) | 6 Years to ≤ 12 Years Age Group: Single Dose 0.10 mg/kg (N=6) | 6 Years to ≤ 12 Years Age Group: Single Dose 0.20 mg/kg (N=7) | 2 Years to < 6 Years Age Group: Single Dose 0.05 mg/kg (N=7) | 2 Years to < 6 Years Age Group: Single Dose 0.10 mg/kg (N=6) | 2 Years to < 6 Years Age Group: Single Dose 0.20 mg/kg (N=6) | 0 to < 2 Years Age Group: Single Dose 0.05 mg/kg (N=7) | 6 Years to ≤ 12 Years Age Group: Multiple Dose 0.20 mg/kg (N=10) | 2 Years to < 6 Years Age Group: Multiple Dose 0.20 mg/kg (N=6)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 6 Years to ≤ 12 Years Age Group: Single Dose 0.05 mg/kg (N=6) | 6 Years to ≤ 12 Years Age Group: Single Dose 0.10 mg/kg (N=6) | 6 Years to ≤ 12 Years Age Group: Single Dose 0.20 mg/kg (N=7) | 2 Years to < 6 Years Age Group: Single Dose 0.05 mg/kg (N=7) | 2 Years to < 6 Years Age Group: Single Dose 0.10 mg/kg (N=6) | 2 Years to < 6 Years Age Group: Single Dose 0.20 mg/kg (N=6) | 0 to < 2 Years Age Group: Single Dose 0.05 mg/kg (N=7) | 6 Years to ≤ 12 Years Age Group: Multiple Dose 0.20 mg/kg (N=10) | 2 Years to < 6 Years Age Group: Multiple Dose 0.20 mg/kg (N=6)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0/2 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0/0 (0) | 0/2 (0)
Procedural anxiety (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Face oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (6) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Clostridium test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incisional drainage (Surgical and medical procedures) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enuresis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This post marketing study was required by the FDA. Endo Pharmaceuticals Inc. no longer promotes opioids and no longer markets Opana® ER.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-08-21): https://cdn.clinicaltrials.gov/large-docs/52/NCT01210352/Prot_SAP_000.pdf